

# The Effect of Eight-week Specific Core Training on Core Stability, Balances and Jumps in young Rhythmic Gymnasts

**Doctorate: Cristina Cabrejas Mata** 

Tutors: Mònica Solana, Jose Morales

Directors: Mònica Solana, Jose Morales

Departament: Ciències de l'activitat física i l'Esport

Date: 30-04-2018

University of Psychology, Education and Sports Science Ramon Llull, Blanquerna.



# INFORMED CONSENT FORM

I, who will sign, as the participant's mother, father or guardian, confirm that (please tick the appropriate box):

| 1. | . I have read and understood the information about the project: "The Effect of Eight-week | | |
|---|---|---|---|
| | Specific Core Training on Core Stability, Balances and Jumps in Young Rhythmic | | |
| | Gymnasts ", explained in the informative document dated | | |
| 2. | I have had the opportunity to ask questions about participation in this project | | |
| 3. | As a parent, guardian or | guardian of the minor partici | pant I agree that (name) |
| | wi | ll voluntarily participate in this pro | oject. |
| 4. | I know that the participant of | can withdraw at any time without | giving any explanation and |
| | will not be penalized for with | drawing or questioned for the reas | son she is withdrawing. |
| 5. | Confidentiality processes have | re been clearly explained. | 1 |
| 6. | Research data, publications a | nd storage of this data have been e | explained. |
| 7. | I understand that other resea | archers will have access to this da | ata, as long as they agree to |
| | preserve the confidentiality of | of the data and also if they agree | to the terms specified in this |
| | form. | | |
| 8. | I, as a parent, guardian, in | agreement with the researcher, | agree to sign and date this |
| | consent form. | | |
| Par | ticipant: | | |
| Name of participant | | Signature | Date |
| Mot | ther, father or guardian: | | |
| Name of mother, father or guardian | | Signature | Date |
| Res | earcher: | | |



### INFORMED CONSENT

| I, | , | father, | mother | or | legal |
|---------------------------------------|------|---------|--------|----|-------|
| guardian of | with | ID | | | , |
| acting in my own name and interest. I | | | | | |

### **DECLARE THAT:**

I have received information about the project "The Effect of Eight-week Specific Core Training on Core Stability, Balances and Jumps in Young Rhythmic Gymnasts" from which I have submitted an information document attached to this consent form and for which my participation is requested. I have understood its meaning, my doubts have been clarified and the actions that will derive from it have been exposed to me. I have been informed of all aspects related to the confidentiality and protection of data regarding the management of personal data involved in the project and the guarantees taken in compliance with Law 15/1999 on the Protection of Personal Data.

My collaboration in the project is entirely voluntary and I have the right to withdraw from it at any time, revoking this consent, without this withdrawal can negatively affect my person in any way. In case of withdrawal, I have the right to have my data deleted from the study file. For all of the above.

## I GIVE MY CONSENT TO:

- 1. Participate in the project "The Effect of Eight-week Specific Core Training on Core Stability, Balances and Jumps in Young Rhythmic Gymnasts".
- 2. That the SAFE research team and the student, Cristina Cabrejas Mata as principal investigator, can manage my personal data and disseminate the information generated by this project. It is guaranteed that my identity and privacy will be preserved at all times, with the guarantees established in Law 15/1999 on data protection and complementary regulations.
- 3. That the SAFE team keep all records made about me in electronic form, with the guarantees and deadlines legally provided, if established, and in the absence of legal provision, for the time necessary to fulfill the functions of the project for which the data were collected.

| In Barcelona on | of2018 | |
|-----------------|----------------------------|------------------------|
| Signatures: | | |
| Participant | Mother, father or guardian | Principal Investigator |